CLINICAL TRIAL: NCT06791434
Title: Investigating Dry Needling As an Add-on Therapy to Conventional Treatment for Myofascial Low Back Pain: a Randomized Controlled Trial
Brief Title: Assessing the Benefits of Dry Needling for Low Back Pain When Combined with Regular Treatment
Acronym: DryNATiMP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Vishwanath Karad MIT World Peace University (Other)
Responsible Party: Principal Investigator, Deshbandhu Pachauri, Principal Investigator, Dr. Vishwanath Karad MIT World Peace University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MITWPU-CS-01
Record Dates: First submitted 2024-12-31; First posted 2025-01-24 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Dry Needling; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Treatment (CT) Group (Active Comparator): Also known as Control group. In this group, patients to follow prescribed pharmacotherapy (Fixed Dose Combination "Etoshine MR" tablets BID) daily for first 2 weeks and prescribed physiotherapy daily until Day 168.
  Interventions: Drug: Fixed Dose Combination "Etoshine MR" tablets; Other: Physiotherapy
- Conventional Treatment + Dry Needling (CT+DN) Group (Experimental): Also known as Add-on group. In this group, in addition to the treatment prescribed for the CT group, patients to also receive 5 dry needling sessions scheduled on Day 0, 3, 7, 10, and 14.
  Interventions: Drug: Fixed Dose Combination "Etoshine MR" tablets; Procedure: Dry needling; Other: Physiotherapy

INTERVENTIONS:
Drug: Fixed Dose Combination "Etoshine MR" tablets — Composition per tablet: Etoricoxib 60 mg + Thiocolchicoside 4 mg
Procedure: Dry needling — Thin needle insertion
  Arms: Conventional Treatment + Dry Needling (CT+DN) Group
Other: Physiotherapy — Exercises

SUMMARY:
The proposed clinical study aims to evaluate the effectiveness and safety of adding Dry Needling (DN) to Conventional Treatment (CT) for patients with Myofascial Low Back Pain (MLBP). MLBP is a widespread musculoskeletal condition that causes localized pain, muscle tenderness, and functional limitations, significantly affecting the quality of life and productivity of those affected. Conventional Treatment for MLBP typically combines pharmacotherapy (e.g., NSAIDs, muscle relaxants) and physiotherapy. Dry Needling, an emerging treatment that targets myofascial trigger points with fine needles, has demonstrated promise in relieving pain and improving functional outcomes. However, no study has yet evaluated the combined effects of CT and DN. This randomized, open-label, controlled trial will involve 140 patients (70 per group) and compare the effects of CT alone versus CT combined with DN. The primary objective is to assess the change in pain intensity, while secondary objectives include improvements in pressure pain threshold, range of motion, disability, quality of life, sleep, anxiety, and depression scores.

Safety will also be assessed based on adverse events and vital sign changes. The study will span 24 weeks, with 11 scheduled visits for each participant. Data analysis will be conducted to determine the added benefit of DN as an adjunctive therapy to CT, with the ultimate goal of improving treatment strategies and patient outcomes for MLBP.

ELIGIBILITY:
Inclusion Criteria:

* Subject diagnosed with myofascial low back pain, characterized by the presence of trigger points and localized muscle pain/tenderness
* Subject experiencing myofascial pain symptoms (e.g., muscle pain, tenderness) for at least 3 months
* Subject has a baseline Numeric Pain Rating Scale (NPRS) score of 4 or higher
* Subject has stable medical condition that is not expected to significantly deteriorate during the study period in the opinion of the investigator
* Woman who is postmenopausal for 12 months or less before screening (unless permanently sterilized or using an IUD) must have a negative urine pregnancy test prior to the randomization visit
* Subject is willing to comply with all aspects of the study protocol, including attending scheduled appointments, completing study assessments and adhering to applicable restrictions
* Subject has provided informed consent to participate in the study
* No spine/lumbar surgery in the last 6 months

Exclusion Criteria:

* Subject presenting sharp, shooting pain radiating to lower limbs (associated with tingling and numbness) along with back pain
* Subject with active systemic or local infection(s)
* Subject with bleeding disorder(s) or on anticoagulant medication(s)
* Subject currently experiencing or with a history of psychiatric condition, cognitive impairment, neurological disorder, or other clinically significant disease or abnormality (such as congestive heart failure, uncontrolled hypertension, myocardial infarction, stroke, uncontrolled coronary artery disease, arrhythmias, uncontrolled diabetes, convulsive disorders etc.) which, in the opinion of the investigator, would put the subject at risk through study participation, or would affect the study analyses if the disease exacerbated during the study, or would interfere with their ability to complete the study, or would hinder their ability to understand the study procedures, or would impact their compliance with study assessments or treatment protocols, or would affect pain perception
* Subject with a history of allergy or hypersensitivity to Etoricoxib, Thiocolchicoside or Diclofenac
* Subject with a history of alcohol or substance abuse
* Woman who is pregnant or planning pregnancy during the course of the study
* Subject who is currently participating in or has participated in any other clinical trial within 3 months prior to screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity using Numeric Pain Rating Scale (NPRS) | Screening, Day 0, 3, 7, 10, 14, 28, 56, 84, 168
  Numeric Pain Rating Scale (NPRS) is a widely used, validated tool for assessing pain intensity. Patients are asked to rate their pain on a scale from 0 to 10, with 0 representing no pain and 10 representing the worst possible pain. This simple and reliable scale allows patients to quantify their pain level, aiding clinicians in monitoring pain over time and assessing the effectiveness of treatment interventions.

SECONDARY OUTCOMES:
Change in Pressure Pain Threshold using Algometer | Day 0, 3, 7, 10, 14, 28, 56, 84, 168
  Pressure Pain Threshold (PPT) measurement using an algometer is a quantitative method employed to assess pain sensitivity in individuals with low back pain. During the assessment, pressure applied to the target area (perpendicular to the muscle) using the algometer probe is gradually increased until the sensation changes from pressure to pain. The pressure at which this transition occurs is recorded as the PPT. This objective measure helps evaluate pain sensitivity and tolerance levels in individuals with low back pain, providing valuable insights into the efficacy of treatment interventions.
Change in Range of Motion | Day 0, 3, 7, 10, 14, 28, 56, 84, 168
  Range of Motion (ROM) assessment is a fundamental component in musculoskeletal evaluation. It provides insights into joint mobility, flexibility, and functional limitations.
  Two specific ROM measurements included in this study are as follows:
  1. Fingertip-to-Floor Distance (FTF) in Flexion: The patient bends forward, attempting to reach the floor with their fingertips. A standard measuring tape gauges the distance between the right long finger and the floor.
  2. Lateral Bending ROM: The distance between middle fingertip and floor during lateral bending is measured.
Change in Physical Disability using Salen's Disability Rating Index (DRI) | Day 0, 7, 14, 28, 56, 84, 168
  Disability Rating Index (DRI) is a patient-reported questionnaire that measures physical disability in patients. It was developed in 1994 by Salén et al. DRI questionnaire comprises of 12 items, each measured using a visual analogue scale [VAS (0-100)], where 0 indicates no disability and 100 an inability to perform any activity. The mean of the 12 items provides the overall DRI score. The items are broadly grouped into three distinct sections: (i) questions 1-4, basic activities of daily life: dressing, outdoor walks, climbing stairs, sitting a long time; (ii) questions 5-8, daily physical activities: standing bent over a sink, carrying a bag, making a bed, running; and (iii) questions 9-12, work-related/more vigorous activities: light work, heavy work, lifting heavy objects and participating in exercise/sports.
Change in Pain and Sleep using Pain and Sleep Questionnaire (PSQ-3) | Day 0, 7, 14, 28, 56, 84, 168
  The Pain and Sleep Questionnaire (PSQ-3) is a concise tool designed to evaluate the influence of pain on sleep quality. Each of the 3 items is scored individually on a 100 mm Visual Analog Scale (VAS), ranging from 0 (representing 'never') to 100 (indicating 'always'). The total score is obtained by summing up the scores of all three items, providing a comprehensive measure of the impact of pain on sleep quality. By quantifying the frequency of sleep disturbances attributed to pain, the PSQ-3 provides valuable insights into the intricate relationship between pain and sleep, crucial for assessing the holistic impact of myofascial low back pain on patients' well-being.
Change in Quality of Life Scale Score using Burckhardt's Quality of Life Scale (QOLS) | Day 0, 7, 14, 28, 56, 84, 168
  Burckhardt's Quality of Life Scale (QOLS) is a self-reported measure assessing overall quality of life across physical, psychological, and social domains. It comprises of 16 items related to life satisfaction, including health, relationships, and daily activities. Participants rate each item, providing insights into their perceived well-being. Each item is scored on a Likert-type scale ranging from 7 to 1, where 7 ="Delighted" to 1 = "Terrible". The QOLS offers a comprehensive assessment, valuable for evaluating the impact of health conditions like myofascial low back pain on quality of life. Total score is obtained by adding up the score on each item. Range of the total score: 16-112. Higher score indicates better quality of life.
Change in Patients Impression using Patients' Global Impression of Change (PGI-C) Scale | Day 3, 7, 14, 28, 56, 84, 168
  Patients' Global Impression of Change (PGI-C) scale allows participants to subjectively assess their overall improvement or worsening of back pain symptoms since the start of the study. It consists of seven options ranging from "Very Much Improved" to "Very Much Worse." The PGI-C scale provides valuable insights into participants' perceptions of the effectiveness of the treatment.
Change in Severity of Anxiety and Depression Symptoms using Hospital Anxiety and Depression Scale (HADS) | Day 0, 7, 14, 28, 56, 84, 168
  Hospital Anxiety and Depression Scale (HADS) is a widely used self-assessment tool designed to measure the severity of anxiety and depression symptoms in individuals with physical health conditions. It consists of 14 items, with seven items each assessing anxiety and depression separately. Respondents rate their feelings over the past week using the respective scores which range from 0 to 3. Higher the score out of 21, higher the severity of anxiety/depression. Monitoring the changes in anxiety and depression scores throughout the study can provide valuable data on the impact of treatment on patients' mental health.

CONTACTS AND LOCATIONS:
Locations (1):
- Sigma Spine and Pain Clinic, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hong CZ. Treatment of myofascial pain syndrome. Curr Pain Headache Rep. 2006 Oct;10(5):345-9. doi: 10.1007/s11916-006-0058-3. PMID 16945250
- [Background] Kalichman L, Vulfsons S. Dry needling in the management of musculoskeletal pain. J Am Board Fam Med. 2010 Sep-Oct;23(5):640-6. doi: 10.3122/jabfm.2010.05.090296. PMID 20823359